CLINICAL TRIAL: NCT04920409
Title: Effect of an Antiinflammatory Diet on Postprandial Gene Expression of Mononuclear Cells of Adult Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Caldas (Other)
Collaborators: Universidad Libre (Unknown); Clínica Comfamiliar Risaralda (Unknown)
Responsible Party: Principal Investigator, Diana M Munoz, Principal investigator, Universidad de Caldas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0406716
Record Dates: First submitted 2021-05-25; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Obesity; Diet; Postprandial state; Gene expression; Inflammation; Lipemia; Insulinemia
MeSH Terms: conditions — Obesity; Inflammation; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAWGT Diet (Experimental): Composed of fruit, avocado, whole grains and trout
  Interventions: Other: FAWGT diet
- Usual diet (UD) (Active Comparator): Based on the food which the participants usually consumed prior to the study in their normal lifestyle.
  Interventions: Other: Usual diet (UD)

INTERVENTIONS:
Other: FAWGT diet — Composed of 15% protein, 55% CH and 30% fat of which < 10% was SFA, 14% MUFA and 6% PUFA in the overall total caloric content.
  Arms: FAWGT Diet
Other: Usual diet (UD) — Consisted of 16% protein, 54% carbohydrates (CH) and 30% fat of which 15% was saturated fat (SFA), 10% monounsaturated fat (MUFA) and 5% polyunsaturated fat (PUFA)in relation to the total caloric content
  Arms: Usual diet (UD)

SUMMARY:
Obesity is one of the major health problems worldwide. The consumption of healthy-dietary patterns can be difficult in some countries due to the availability of certain foods. Suggestion of alternative foods could be a necessity. The purpose of this study was to evaluate the effect of a dietary pattern consisting of fruit, avocado, whole-grains and trout (FAWGT) on postprandial gene expression, insulinemia and lipemia in Colombian obese people.

DETAILED DESCRIPTION:
A randomized controlled crossover study was conducted. Volunteers underwent to two dietary models for 8 weeks each, including a 2 weeks washout diet between them. The order in which they started the interventions was randomized following a computerized assignment list using Excel software (Microsoft Office 2015, Excel 2013).

The primary endpoint was the postprandial gene expression of nuclear factor kappa B subunit 1 (NFKB1) gene. Based on previous studies , 20 individuals had to be studied to detect a 0.2 difference in the expression of the NKKB1 gene between diets with 0.05 significance level and 80 percentage power (type II error Z 0.2), assuming a 10 percentage drop-out rate.

The recruitment of participants was carried out according to the following steps:

1. Review of clinical histories of patients diagnosed with obesity, according to their Body Mass Index, ascribed to the chronic non-communicable diseases program of the Clinica Comfamiliar Risaralda in the city of Pereira Colombia.
2. Telephone call to invite the participants who met the inclusion criteria to participate in the study.
3. Appointment prior to the start of the study to take a blood sample to corroborate the inclusion criteria. With this sample the following tests were performed: blood glucose, lipid profile, thyroid stimulating hormone (TSH), C-reactive protein ( and complete blood count.

This process was carried out by personnel not involved in the research. The results obtained were compared with the clinical history.

The diets followed during the intervention periods were: (1) a diet consisting mainly of the consumption of fruit, avocado and other vegetables, whole grains and trout typical of the colombian coffee region (FAWGT) (experimental diet), and (2) the usual diet consumed by the participants in their normal lifestyle (UD).

At the beginning of the dietary intervention period, each participant was given an individualized food guide containing the suggested food group and portions, with a wide variety of foods allowed for greater adherence to the diet. In addition, specific times for consumption of the foods and precise instructions for the dietary intervention were given. In addition, the subjects were given a talk advising them how to quantify the portions, which would later be converted into grams according to the procedure described

The food portions were standardized with all the participants using synthetic models, adapted according to the Colombian nutritional guidelines, so that they could provide a more accurate report of the portions consumed during the intervention. In addition, a postprandial studies were carried out at the beginning of the study (pre-intervention) and another after 8 weeks of dietary intervention (post-intervention).

The participants were given an appointment at the health center at 7.00 am, after at least 12 hours of fasting and a 5 day abstinence from alcohol. They consumed a breakfast based on the same composition of the diet in which they were randomized for the dietary intervention period. The blood samples were obtained by veni-puncture at baseline and 4 hours after breakfast. During the postprandial period, the participants did not consume any more food, although they were allowed to drink water. The breakfasts were composed of the following foods: FAWGT diet; whole-grain arepa (with unrefined corn flour), cheese, oats, granadilla, mango, linseed, nuts, almonds, peanuts and yogurt. Usual diet; egg, cheese, butter, whole milk, traditional white arepa (with re-fined corn flour), traditional buñuelo (made from wheat flour with cheese), coffee and sugar.

Before starting the dietary intervention period (Pre-intervention), at the midpoint of the study (week 4) and at the end (week 8), all the participants completed three 24-hour recalls (2 non-consecutive weekdays and one weekend day) to obtain information about food, ingredients and preparations consumed in the same units of measurement (grams).

In addition, a weekly telephone call was made to answer any questions relating to the diet (recipes, menu and quantities) and to motivate adherence to the assigned dietary model.

Moreover, in week four of each intervention, the participants attended the hospital for an interview with the main researcher in order to take anthropometric measurements, evaluate the follow-up of the dietary instructions and answer any questions that may have arisen during the intervention, and motivate them to continue with the study. To collect the information on food consumption, formats and questionnaires previously published by the research group were used.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Body mass index (BMI) ≥ 30 Kg/m^2.
* Clinical: hypertensive and dyslipidemic participants.

Exclusion Criteria:

* Age < 40 or > 65 years
* Patients unable to follow a protocol.
* Psychiatric diseases
* Renal Insufficiency
* Chronic Hepatopathy
* Active Malignancy
* Chronic obstructive pulmonary disease
* Diseases of the digestive tract Endocrine disorders
* Smokers.
* Regular alcohol consumers.
* Participants who were in weight reduction programs
* Prescribed hypolipidaemic medication
* Prescribed anti-inflammatory medication
* Kidney or liver dysfunction.
* Diabetes or other endocrine disorders.
* Chronic inflammatory conditions.
* Patients participating in other Clinical trials (in the enrollment moment or 30 days prior).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Relative expression of the NFKB1 gene | 8 weeks
  RNA extraction from mononuclear cells, reverse transcription and DNA amplification in fasting and postprandial state.
Relative expression of the Interleukin 6 (IL6) gene | 8 weeks
  RNA extraction from mononuclear cells, reverse transcription and DNA amplification in fasting and postprandial state.
Relative expression of the tumoral necrosis factor (TNF) gene | 8 weeks
  RNA extraction from mononuclear cells, reverse transcription and DNA amplification in fasting and postprandial state.
Relative expression of the Interleukin 1 B (IL1B) gene | 8 weeks
  RNA extraction from mononuclear cells, reverse transcription and DNA amplification in fasting and postprandial state..
Relative expression of the matrix metallopeptidase 9 (MMP)) gene | 8 weeks
  RNA extraction from mononuclear cells, reverse transcription and DNA amplification in fasting and postprandial state.
Relative expression of the nuclear factor, erythroid 2 like 2 (NFE2L2) gene | 8 weeks
  RNA extraction from mononuclear cells, reverse transcription and DNA amplification.

SECONDARY OUTCOMES:
Change from baseline of the gut microbiota | 8 weeks
  Stool deoxyribonucleic acid (DNA) extraction, library construction, sequencing and bioinformatic analysis.
Change from baseline of DNA methylation pattern | 8 weeks
  Whole blood DNA extraction and Enzyme-Linked ImmunoSorbent Assay (ELISA)
Triglycerides | 8 weeks
  Influence of diet on postprandial trygliceride
Insulin | 8 weeks
  Influence of diet on postprandial insulinemia
Total Cholesterol | 8 weeks
  Influence of diet on postprandial total Cholesterol
LDL Cholesterol | 8 weeks
  Influence of diet on postprandial LDL Cholesterol
HDL Cholesterol | 8 weeks
  Influence of diet on postprandial HDL Cholesterol
VLDL Cholesterol | 8 weeks
  Influence of diet on postprandial VLDL Cholesterol
C-reactive protein (CRP) | 8 weeks
  Influence of diet on postprandial CRP

CONTACTS AND LOCATIONS:
Overall Officials: Clara H Gonzalez Correa, Doctor, Study Director — Universidad de Caldas; Diana M Muñoz, PhD student, Principal Investigator — Universidad de Caldas; Oriol A Rangel Zuñiga, Postdoctor, Principal Investigator — Instituto Maimonides de Investigación Biomédica de Córdoba; Antonio Camargo, Postdoctor, Principal Investigator — Instituto Maimonides de Investigacion Biomedica de Cordoba; Elcy Y Astudillo Muñoz, Doctor, Study Chair — Universidad Libre; Gloria L Porras Hurtado, Postdoctor, Study Chair — Clinica Comfamiliar Risaralda; Maite Sanchez Giraldo, PhD student, Study Chair — Instituto Maimonides de Investigación Biomedica de Cordoba
Locations (1):
- Clinica Comfamiliar Risaralda, Pereira, Risaralda Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurt RT, Kulisek C, Buchanan LA, McClave SA. The obesity epidemic: challenges, health initiatives, and implications for gastroenterologists. Gastroenterol Hepatol (N Y). 2010 Dec;6(12):780-92. PMID 21301632
- [Background] Frigolet ME, Dong-Hoon K, Canizales-Quinteros S, Gutierrez-Aguilar R. Obesity, adipose tissue, and bariatric surgery. Bol Med Hosp Infant Mex. 2020;77(1):3-14. doi: 10.24875/BMHIM.19000115. PMID 32115585
- [Background] Fernemark H, Jaredsson C, Bunjaku B, Rosenqvist U, Nystrom FH, Guldbrand H. A randomized cross-over trial of the postprandial effects of three different diets in patients with type 2 diabetes. PLoS One. 2013 Nov 27;8(11):e79324. doi: 10.1371/journal.pone.0079324. eCollection 2013. PMID 24312178
- [Background] Koch W. Dietary Polyphenols-Important Non-Nutrients in the Prevention of Chronic Noncommunicable Diseases. A Systematic Review. Nutrients. 2019 May 9;11(5):1039. doi: 10.3390/nu11051039. PMID 31075905
- [Background] Lopez-Miranda J, Williams C, Lairon D. Dietary, physiological, genetic and pathological influences on postprandial lipid metabolism. Br J Nutr. 2007 Sep;98(3):458-73. doi: 10.1017/S000711450774268X. PMID 17705891
- [Background] Perez-Martinez P, Ordovas JM, Garcia-Rios A, Delgado-Lista J, Delgado-Casado N, Cruz-Teno C, Camargo A, Yubero-Serrano EM, Rodriguez F, Perez-Jimenez F, Lopez-Miranda J. Consumption of diets with different type of fat influences triacylglycerols-rich lipoproteins particle number and size during the postprandial state. Nutr Metab Cardiovasc Dis. 2011 Jan;21(1):39-45. doi: 10.1016/j.numecd.2009.07.008. Epub 2009 Oct 9. PMID 19819118
- [Background] Uusitupa M, Hermansen K, Savolainen MJ, Schwab U, Kolehmainen M, Brader L, Mortensen LS, Cloetens L, Johansson-Persson A, Onning G, Landin-Olsson M, Herzig KH, Hukkanen J, Rosqvist F, Iggman D, Paananen J, Pulkki KJ, Siloaho M, Dragsted L, Barri T, Overvad K, Bach Knudsen KE, Hedemann MS, Arner P, Dahlman I, Borge GI, Baardseth P, Ulven SM, Gunnarsdottir I, Jonsdottir S, Thorsdottir I, Oresic M, Poutanen KS, Riserus U, Akesson B. Effects of an isocaloric healthy Nordic diet on insulin sensitivity, lipid profile and inflammation markers in metabolic syndrome -- a randomized study (SYSDIET). J Intern Med. 2013 Jul;274(1):52-66. doi: 10.1111/joim.12044. Epub 2013 Mar 2. PMID 23398528
- [Background] Gomez-Marin B, Gomez-Delgado F, Lopez-Moreno J, Alcala-Diaz JF, Jimenez-Lucena R, Torres-Pena JD, Garcia-Rios A, Ortiz-Morales AM, Yubero-Serrano EM, Del Mar Malagon M, Lai CQ, Delgado-Lista J, Ordovas JM, Lopez-Miranda J, Perez-Martinez P. Long-term consumption of a Mediterranean diet improves postprandial lipemia in patients with type 2 diabetes: the Cordioprev randomized trial. Am J Clin Nutr. 2018 Nov 1;108(5):963-970. doi: 10.1093/ajcn/nqy144. PMID 30475968